CLINICAL TRIAL: NCT05878743
Title: A Survivor Researcher-led Qualitative Mixed Methods Realist Evaluation of Safety Planning: a Recovery-orientated Mental Health Risk Management Intervention.
Brief Title: A Qualitative Mixed Methods Realist Evaluation of Safety Planning
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 293012
Record Dates: First submitted 2023-05-19; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Risk Behavior, Health
MeSH Terms: conditions — Health Risk Behaviors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Safety Planning a recovery-orientated mental health risk management intervention — Developing the skills to manage risks associated with mental health difficulties in ways which increase personal recovery for individuals.

SUMMARY:
Safety Planning is a recovery-orientated approach to risk management within mental health context. This study wants to answer the question 'how, why, for whom and it what circumstances does safety planning work? It will do this by carrying out a realist evaluation to identify programme theories by conducting a three phase study, reviewing materials of a Safety Planning training course, interviewing service users, carers and mental health professionals who have attended the training course, and/or use safety planning tools and techniques, adopting theory from existing literature and adding evaluator's insider knowledge. This data will be used to describe programme theory of safety planning that can be applied across diverse mental health settings, including NHS inpatient and community, and is designed to be adopted across different contexts. It will use a realist methodology to understand how safety planning works to develop the skills needed to manage risks associated with mental health difficulties in ways which increase an individual's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Service user participants - must have direct lived experience of managing safety from risks associated with their mental health difficulties / have attended the safety planning recovery college course delivered within Norfolk & Suffolk NHS Foundation Trust (NSFT) / Be accessing a service from NSFT and have an identified care team, lead care professional and/or know how to access help and support.

Carer participants - have cared for someone who lived with risks associated with their mental health difficulties / have attended the safety planning recovery college course delivered by NSFT / know how to access emotional support should they require it during the study Mental health professionals - have either a) supported people in a professional capacity to manage risks associated with mental health difficulties, b) attended either the safety planning recovery college course (NSFT) OR a version of safety planning training delivered within NSFT c) have some responsibility for safety planning and risk management within the trust. MUST HAVE knowledge of how to access staff wellbeing and support systems for emotional support should they require it during the study.

Exclusion Criteria:

* People under 16 years of age / people who are unable to communicate in English / people with no access to computer, internet or basic IT skills /

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Mental health service users accessing a service from Norfolk & Suffolk NHS Foundation Trust, Carers (family members, friends) of someone accessing a service from NSFT and Mental Health practitioners.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-05-16 (Estimated)

PRIMARY OUTCOMES:
Formal theory described which explains how, why, for whom and in what circumstances safety planning works. | two years

IPD SHARING:
Plan to Share IPD: Undecided